CLINICAL TRIAL: NCT03584646
Title: Development and Testing of a Prehabilitation Intervention to Maximize Early Recovery (PRIMER) in Liver Transplantation
Brief Title: Prehabilitation Intervention to Maximize Early Recovery (PRIMER) in Liver Transplantation
Acronym: PRIMER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Marina Serper, MD, MS, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 828669
Record Dates: First submitted 2018-02-01; First posted 2018-07-12 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Liver Diseases; End Stage Liver Disease; Frailty
Keywords: liver transplantation; malnutrition; exercise; prehabilitation; nutrition; sarcopenia
MeSH Terms: conditions — Liver Diseases; End Stage Liver Disease; Frailty; Malnutrition; Motor Activity; Sarcopenia

STUDY DESIGN:
Intervention Model Description: The investigator will conduct a patient-randomized, two-arm pilot study of 38 participants with a predicted attrition rate of 20% resulting in 30 total participants; n=10 in Arm 1 and n=20 in Arm 2. Arm 1 will serve as the control arm and Arm 2 will serve as the intervention arm.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Control Arm (Experimental): Usual care, nutrition and exercise counseling at baseline, use of the Nokia GO wearable step tracker device and end-of-study assessment at the end of the 14-week study period. Participants will receive the Nokia GO wearable step tracker to monitor daily step counts, but they will not be provided with personalized walking goals or automated feedback on goal attainment via text message.
  Interventions: Device: Nokia GO Wearable StepTracker
- Arm 2 - Intervention arm (Experimental): Physical activity program supported by financial incentives for meeting walking goals and participating in weekly check-in appointments with study team members via telephone calls. Participants in the intervention arm will also receive twice-daily medication reminders via bidirectional text messages to promote medication adherence. Participants in Arm 2 will also receive personalized nutrition and exercise counseling, daily feedback on step counts via the Nokia GO wearable step tracker and their smartphones, and an end-of-study assessment.
  Interventions: Device: Nokia GO Wearable StepTracker; Other: Medication Reminder; Other: Weekly Check-in appointment with study team or provider

INTERVENTIONS:
Device: Nokia GO Wearable StepTracker — All participants will be provided with a Nokia GO step tracker to monitor daily step counts. The device is not subject to FDA regulation.
Other: Medication Reminder — Medication reminders are sent to participants in Arm 2 on a daily basis.
  Arms: Arm 2 - Intervention arm
Other: Weekly Check-in appointment with study team or provider — Virtual meeting or telephone call between participants and study team to assess study involvement, adherence to procedures, and following of medical care recommendations.
  Arms: Arm 2 - Intervention arm

SUMMARY:
This is a single center, 2-arm, patient-randomized study evaluating the feasibility and potential efficacy of the PRIMER intervention in improving physical function and reducing frailty in adult Liver Transplant candidates. The intervention will consist of a patient-tailored prehabilitation program designed to reduce frailty, improve physical function and nutritional status, and optimize pre- and post-transplant outcomes.

DETAILED DESCRIPTION:
The investigator will pilot-test a two-arm, randomized trial of a prehabilitation intervention in 38 pre-liver transplant patients with End Stage Liver Disease (ESLD). The investigator estimates an attrition rate of 20%, resulting n=30 participants; 10 participants in Arm 1 (control arm) and 20 participants in Arm 2 (intervention arm). To be eligible, patients must be waitlisted or "Penn-Ready" with a MELD-Na less than or equal to 25, English-speaking, able to safely participant in an exercise program, have a smartphone, and be identified as frail. The purpose of this trial is to develop and implement a program of medical optimization, physical activity, and nutrition recommendations specifically tailored to ESLD and designed to reduce frailty, improve physical function, and optimize pre- and post-transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be wait-listed, in transplant evaluation, or "Penn Ready" with a MELD-Na score less than or equal to 25;
2. Patients must be English speaking and own/use a smartphone and cognitively able to consent;
3. Patient and physician feel that individual can safely participate in an exercise program;
4. Meeting at least one 'at risk' criterion for impaired physical performance, frailty, or malnutrition (by SPPB, abPG-SG, dynamometer measured grip strength), or physical deconditioning as determined by physical therapist, or treating clinician.

Exclusion Criteria:

1. The patient is unable to provide informed consent;
2. The patient has been hospitalized within the last 30 days;
3. A score of 0-3 points on the SPPB assessment indicating inability to participate in a physical activity program or a score of 12 in the absence of frailty or malnutrition (indicating low risk for poor physical or performance or malnutrition);
4. The patient is at risk for falling as defined by clinician assessment results or if the patient states that he/she has a history of falling (record of a fall(s) in the past 30 days);
5. The patient is already enrolled in a financial incentive-based exercise program using a wearable device;
6. Any other medical conditions that would prohibit participation in a physical activity program as determined by transplant clinicians or severe vision, hearing, or mobility impairment precluding participation.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Intervention | 14 weeks
  Feasibility of the intervention will be evaluated by the percentage of patients that complete the study intervention.
Acceptability of the Intervention | 14 weeks
  Acceptability will be measured using a patient satisfaction questionnaire upon study completion.

SECONDARY OUTCOMES:
Performance on the Short Physical Performance Battery (SPPB) | 14 weeks
  The SPPB is a simple test to measure lower extremity function using tasks that mimic daily activities. The SPPB examines three areas of lower extremity function; static balance, gait speed, and getting in and out of a chair. Static balance is measured in units of time (seconds) and patients are timed holding 3 different stances. Gait speed is measured in time (seconds) to walk 4 meters. Chair sits are measured as the time (seconds) it takes to get up and out of a chair 5 times without using one's arms to assist the exercise. Collectively, the three tests are used to generate a total score (0-12) that reflects a patient's frailty (score of 0) or lack of frailty (score of 12).
Grip strength | 14 weeks
  Grip strength will be measured using a digital hand dynamometer and the unit of measure is kilograms.
Grip strength level relative to BMI | 14 weeks
  Body Mass Index (BMI) will be calculated using height in inches and weight in pounds and reported as 'kg/m^2'. Grip strength will be compared to BMI and a 'BMI-adjusted' grip strength level will be reported using established 'kilogram to BMI ratio' standards.
Body composition/BIA | 14 weeks
  Bioelectrical impedance analysis will be completed using the Bodystat Quadscan 4000, which is a multi-frequency body composition analyzer. Body fat percentage (%) will be compared to lean body mass percentage and total body water percentage to assess sarcopenia and nutritional status.

OTHER OUTCOMES:
Clinical Outcomes from Medical Record Review - Liver Transplant listing | 12 months
  A medical record review will be conducted at the end of the study to review clinical outcomes, liver transplant listing date and occurrence will be assessed.
Clinical Outcomes from Medical Record Review - Liver Transplantation | 12 months
  A medical record review will be conducted at the end of the study to review clinical outcomes, date and occurrence liver transplantation will be assessed.
Clinical Outcomes from Medical Record Review - Death | 12 months
  A medical record review will be conducted at the end of the study to review clinical outcomes, occurrence and/or date of death will be assessed.
Clinical Outcomes from Medical Record Review - Hospitalization | 12 months
  A medical record review will be conducted at the end of the study to review clinical outcomes, number of admissions/hospitalizations will be assessed.
Clinical Outcomes from Medical Record Review - Removal from Liver Transplant List | 12 months
  A medical record review will be conducted at the end of the study to review clinical outcomes, occurrence and date of removal from the liver transplant list will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No